CLINICAL TRIAL: NCT02019407
Title: Prospective Randomized Study on Clinical Effectiveness of Carvo-Tricuspid Isthmus Block in Patients With Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2013-0639
Record Dates: First submitted 2013-12-06; First posted 2013-12-24 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial flutter; catheter ablation; cavo-tricuspid isthmus block
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTI group (Experimental): CTI(Cavo-Tricuspid Isthmus)
  Interventions: Procedure: PVI, CTI block
- Non CTI group (Placebo Comparator): Non CTI (Cavo-Tricuspid Isthmus)
  Interventions: Procedure: PVI

INTERVENTIONS:
Procedure: PVI, CTI block — * PVI (pulmonary isolation)
  * Catheter ablation of cavo-tricuspid isthmus line for treatment of atrial fibrillation
  Catheter is inserted into inferior venacava (IVC) and right atrium (RA) via femoral vein. And the procedure is to block bidirectionally between inferior venacava (IVC) and the annulus of tricuspid valve (TV) by using electrical energy of catheter tip.
  Other Names: radiofrequency catheter ablation (RFCA), Catheter ablation of cavo-tricuspid isthmus line for treatment of atrial flutter
  Arms: CTI group
Procedure: PVI — PVI (pulmonary isolation)
  Arms: Non CTI group

SUMMARY:
Prospective Randomized Study on Clinical Effectiveness of Carvo-Tricuspid Isthmus (CTI) Block in Patients with Paroxysmal Atrial Fibrillation (PAF) will be performed. Study will be composed with two arms including 4 pulmonary vein isolation and pulmonary vein isolation with CTI block. After that all patients will be followed up by HRS(Heart Rhythm Society) 2010 expert consensus guideline.

ELIGIBILITY:
Inclusion Criteria:

* patients with documented AF
* Drug refractory AF
* Non-valvular AF
* No structural cardiac disease
* No intracardiac thrombi in cardiac CT and TEE

Exclusion Criteria:

* permanent AF refractory to electrical cardioversion
* LA size >55 mm as measured by echocardiography
* AF with valvular disease
* associated structural heart disease other than left ventricular hypertrophy
* prior AF ablation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-01; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial fibrillation (AF free survival) | 3 month after catheter ablation
  clinical recurrence of AF after catheter ablation

CONTACTS AND LOCATIONS:
Locations (1):
- ivision of Cardiology, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Mohanty S, Mohanty P, Di Biase L, Bai R, Santangeli P, Casella M, Dello Russo A, Tondo C, Themistoclakis S, Raviele A, Rossillo A, Corrado A, Pelargonio G, Forleo G, Natale A. Results from a single-blind, randomized study comparing the impact of different ablation approaches on long-term procedure outcome in coexistent atrial fibrillation and flutter (APPROVAL). Circulation. 2013 May 7;127(18):1853-60. doi: 10.1161/CIRCULATIONAHA.113.001855. Epub 2013 Apr 9. PMID 23572499